CLINICAL TRIAL: NCT01796977
Title: A Prospective, Multi-Center, Randomized, Open Label Controlled Trial Using a Dissolved Oxygen Enriched Dressing in Nipple-sparing Mastectomy
Brief Title: Using A Dissolved Oxygen Enriched Dressing in Nipple-sparing Mastectomy
Acronym: NSM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to enroll in this subject population
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-12-0001
Record Dates: First submitted 2013-01-09; First posted 2013-02-22 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Reconstructive Breast Surgery
Keywords: Nipple-sparing Mastectomy; NSM; Nipple Sparing Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OxyGenesys Dissolved Oxygen Dressing (Active Comparator): OxyGenesys Dissolved Oxygen Dressing is a closed-cell foam wound dressing enriched with gaseous and dissolved oxygen for use in the management of wounds.
  Interventions: Device: OxyGenesys Dissolved Oxygen Dressing
- Standard Gauze Dressing (Placebo Comparator): A sterile 4x4 covered by an adhesive Tegaderm will serve as the comparator for this study.
  Interventions: Device: Standard Gauze Dressing

INTERVENTIONS:
Device: OxyGenesys Dissolved Oxygen Dressing
  Arms: OxyGenesys Dissolved Oxygen Dressing
Device: Standard Gauze Dressing
  Arms: Standard Gauze Dressing

SUMMARY:
This study will evaluate the effect of OxyGenesys Dissolved Oxygen Dressing in wound complication rates of the nipple areolar complex after a nipple sparing mastectomy.

DETAILED DESCRIPTION:
This study will recruit women who are undergoing a bilateral mastectomy for either cancer or a positive BRCA gene. Women will be randomized to a different treatment per breast. One breast will receive the OxyGenesys dressing and the other will receive the standard gauze dressing. The study will evaluate wound complication rates and compare the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to give written consent
* Females >21 years of age
* At least one breast diagnosed with cancer or mastectomy due to a positive BRCA gene mutation test.
* Subject is indicated for bilateral nipple-sparing mastectomy surgery with immediate breast reconstruction
* Subject is able to comply with the study protocol

Exclusion Criteria:

* Primary tumor(s) located within 2cm of the areola margins
* Inability to perform follow up assessments
* Radiation treatment within 30 days of surgery
* Dermabond or other forms of surgical glue is used in the peri-areola region
* Subjects who are known to be allergic to any of the test product(s) or any component of the test product(s)
* Women who are pregnant
* Subjects who have been treated with an investigational drug or device within the past 30 days prior to enrollment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Curd, MS, Study Director — Halyard Health
Locations (7):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Bodyaesthetic, St Louis, Missouri
  - Aesthetic Plastic Surgery, Great Neck, New York
  - Columbia University, New York, New York
  - New York Group, Tarrytown, New York
  - UT Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- OxyGenesys Dissolved Oxygen Dressing and Gauze Dressing: OxyGenesys Dissolved Oxygen Dressing is a closed-cell foam wound dressing enriched with gaseous and dissolved oxygen for use in the management of wounds.
  Standard Gauze Dressing: A sterile 4x4 covered by an adhesive Tegaderm will serve as the comparator for this study.
  Each study participant acted as her own control (one breast of each participant was treated with OxyGenesys, while the other breast was treated with the standard dressing (control)).
Period: Overall Study
Arm/Group | OxyGenesys Dissolved Oxygen Dressing and Gauze Dressing
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- OxyGenesys Dissolved Oxygen Dressing and Gauze Dressing: OxyGenesys Dissolved Oxygen Dressing is a closed-cell foam wound dressing enriched with gaseous and dissolved oxygen for use in the management of wounds.
  Standard Gauze Dressing: A sterile 4x4 covered by an adhesive Tegaderm will serve as the comparator for this study.
  Each study participant was supposed to act as her own control (one breast to be treated with the test article, the other breast with the control article).
Arm/Group | OxyGenesys Dissolved Oxygen Dressing and Gauze Dressing
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.01 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effects of OxyGenesys Dissolved Oxygen Dressing in Wound Complication Rates of the Nipple Areolar Complex Post Nipple-sparing Mastectomy
Description: Wound Complication Rate
Time Frame: 30 days
Population: Each participant acted as her own control - one breast of each participant received the OxyGenesys Dressing, the other breast received the standard dressing.
Measure: Number; unit: breasts
Units Other Than Participants: breasts
Groups:
- OxyGenesys Dissolved Oxygen Dressing: OxyGenesys Dissolved Oxygen Dressing is a closed-cell foam wound dressing enriched with gaseous and dissolved oxygen for use in the management of wounds.
  OxyGenesys Dissolved Oxygen Dressing
- Standard Gauze Dressing: A sterile 4x4 covered by an adhesive Tegaderm will serve as the comparator for this study.
  Standard Gauze Dressing
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Gauze Dressing
Number analyzed (Participants) | 27 | 27
Number analyzed (breasts) | 27 | 27
breasts | 5 | 5

2. Secondary Outcome: To Evaluate Scar Formation 30 Days Post Nipple-sparing Mastectomy
Description: Patient and Observer Scar Assessment Scale - range = 1 - 10. "1" is best condition ("normal skin") and "10" is worst condition ("worst scar imaginable"). The scale is used to assess each of six different wound characteristics, including vascularity, pigmentation, thickness, relief, pliability, and surface area. The means of these combined scores and their respective standard deviations are reported for each study group. The range of the final evaluation score, based on the collective evaluation of each of the six wound characteristics is "6" (if each of the six scores equals "1") to "60" (if each of the six scores equals "10").
Time Frame: 30 days post nipple-sparing mastectomy
Population: Each participant acted as her own control - one breast received OxyGenesys, while the other breast received the standard dressing. Two patients in the OxyGenesys study arm, and one patient in the Control study arm did not provide follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Gauze Dressing
Number analyzed (Participants) | 25 | 26
units on a scale | 19 (13) | 18 (12)

3. Secondary Outcome: To Assess Pain Using the Numerical Rating Scale
Description: Numerical Rating Scale (NRS) - range = 0 - 10. "0" corresponds to "no pain" and "10" indicates "worst pain imaginable". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: 30 days
Population: There is just one NRS value calculated for the indicated time-frame, and thus a comparison between study groups with respect to this outcome was not made. The single NRS value at 30 days is reported here. One patient did not provide follow-up data at this time-point, and thus the total number of participants is 26 instead of 27 for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Available Study Participants: Each study participant was treated with OxyGenesys Dissolved Oxygen Dressing on one breast and standard gauze dressing on the opposite breast.
Arm/Group | All Available Study Participants
Number analyzed (Participants) | 26
units on a scale | 0.27 (0.6)

4. Secondary Outcome: To Evaluate Scar Formation 30 Days Post Nipple-sparing Mastectomy
Description: as for outcome 2
Time Frame: 30 days post nipple-sparing mastectomy
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Gauze Dressing
Number analyzed (Participants) | 25 | 26
units on a scale | 19 [6 to 51] | 18 [6 to 57]

ADVERSE EVENTS:
Arm/Group | OxyGenesys Dissolved Oxygen Dressing | Standard Gauze Dressing
Serious Adverse Events (participants affected / at risk) | 4/27 | 1/27
Other Adverse Events (participants affected / at risk) | 19/27 | 7/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OxyGenesys Dissolved Oxygen Dressing (N=27) | Standard Gauze Dressing (N=27)
wound necrosis (General disorders) | 3 (3) | 0 (0)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
debridgement (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OxyGenesys Dissolved Oxygen Dressing (N=27) | Standard Gauze Dressing (N=27)
epidermolysis (Congenital, familial and genetic disorders) | 3 (3) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
pyrexia (General disorders) | 1 (1) | 1 (1)
pain (General disorders) | 1 (1) | 1 (1)
necrosis (General disorders) | 12 (12) | 2 (2)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
wound infection (Infections and infestations) | 0 (0) | 1 (1)
incision site pruritus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
drain removal (Surgical and medical procedures) | 1 (1) | 0 (0)
seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
debridgement (Surgical and medical procedures) | 0 (0) | 1 (1)
breast hematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
purulent discharge (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less